CLINICAL TRIAL: NCT05835609
Title: Phase I, Open-label, Dose-escalating, Clinical and Pharmacokinetic Study of PM534 Administered Intravenously to Patients With Advanced Solid Tumors
Brief Title: PM534 Administered Intravenously to Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PM534-A-001-22
Record Dates: First submitted 2023-02-07; First posted 2023-04-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Patients With Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM534 (Experimental): Patients will be included in cohorts of a minimum of three or six patients to receive PM534 at successively increasing dose levels.
  Interventions: Drug: PM534

INTERVENTIONS:
Drug: PM534 — PM534 drug product is provided as a powder for concentrate for solution for infusion, is a sterile, preservative-free, lyophilized white cake in a single-dose vial for reconstitution prior to intravenous infusion.

SUMMARY:
The goals of this trial are to identify the dose limiting toxicities, to determine the maximum tolerated dose and the recommended dose of PM534 in patients with advanced solid tumors. All Patients will receive PM534 via intravenous.

DETAILED DESCRIPTION:
This is a prospective, open-label, dose-escalating phase I study in patients with advanced solid tumors. Patients will be included in cohorts of a minimum of three or six patients to receive PM534 at successively increasing dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent, obtained prior to any specific study procedure.
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1
3. Patients must have:

   3.1 Pathologically confirmed diagnosis of advanced solid tumors 3.2 No more than three prior chemotherapy lines.
4. Patients with measurable or non-measurable disease according to the RECIST v.1.1.
5. Recovery to grade ≤1 from drug-related adverse events (AEs) of previous disease treatments, excluding grade 2 alopecia.
6. Laboratory values within seven days prior to first infusion:

   1. Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L, platelet count ≥100 x 10⁹/L and hemoglobin ≥9 g/dL
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x upper limit of normal (ULN).
   3. Total bilirubin ≤ULN (up to 1.5 x ULN for patients with Gilbert's syndrome).
   4. Creatinine clearance ≥30 mL/min or serum creatinine ≤1.5 x ULN.
   5. Serum albumin ≥3 g/dL.
   6. Serum potassium ≥3.5 mmol/L.
   7. Serum magnesium ≥1.6 mg/dL.
7. Wash-out periods:

   1. At least three weeks since the last chemotherapy.
   2. At least four weeks since the last monoclonal antibody (MAb)-containing therapy.
   3. At least two weeks since the last biological/investigational single-agent therapy (excluding MAbs) and/or palliative radiotherapy (RT).
   4. In patients with hormone-sensitive breast cancer progressing while on hormone therapy (except for luteinizing hormone-releasing hormone [LHRH] analogues in pre-menopausal women or megestrol acetate), all other hormonal therapies must be stopped at least one week before study treatment start.
   5. Castrate-resistant prostate cancer (CRPC) patients may continue receiving hormone therapy prior to and during study treatment.
8. Life expectancy ≥3 months

Exclusion Criteria:

1. Concomitant diseases/conditions:

   1. Increased cardiac risk:

      * History of long QT syndrome.
      * Corrected QT interval (QTcF, Fridericia correction) ≥450 msec on screening electrocardiogram (ECG).
      * History of or current ischemic heart disease, including myocardial infarction, stable/unstable angina, coronary arteriography or cardiac stress testing with findings consistent with coronary occlusion or infarction or symptomatic arrhythmia.
      * History of heart failure or left ventricular dysfunction (left ventricular ejection fraction [LVEF] ≤50%) by multiple-gated acquisition scan (MUGA) or echocardiography (ECHO).
      * Clinically significant ECG abnormalities, including any of the following: right bundle branch block with left anterior hemiblock, second (Mobitz II) or third degree atrioventricular block and findings suggestive of ischemic heart disease.
      * Symptomatic arrhythmia.
      * Use of a cardiac pacemaker.
      * History of or current peripheral vascular disease or cerebrovascular disease.
   2. Presence of:

      * Any grade of peripheral neuropathy (any etiology) at study entry.
      * Prior history of grade ≥ 2 peripheral neuropathy due to any chemotherapeutic or investigational agent.
      * Clinical or radiological signs of subocclusion/bowel obstruction.
   3. Active infection requiring systemic treatment.
   4. Known human immunodeficiency virus (HIV) or known hepatitis C virus (HCV) infection or active hepatitis B.
   5. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study
2. Symptomatic, steroid-requiring, central nervous system (CNS) disease.
3. Patients with carcinomatous meningitis.
4. Prior bone marrow or stem cell transplantation.
5. Current treatment with colchicine.
6. Use of (strong or moderate) inhibitors or strong inducers of CYP3A4 activity within two weeks prior to the first infusion of PM534
7. Known hypersensitivity to any of the components of the drug product.
8. Limitation of the patient's ability to comply with the treatment or to follow the protocol procedures.
9. Women who are pregnant or breast feeding and fertile patients (men and women) who are not using an effective method of contraception
10. Patients with pulmonary lymphangitis.
11. Use of medications with known risk of inducing torsades de pointes (TdP) within five half-lives prior to the first infusion of PM534

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Determination of the Maximum Tolerated Dose and the Recommended Dose | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  A fully evaluable patient is a patient evaluable for the primary objective (i.e., determination of the MTD and the RD).

SECONDARY OUTCOMES:
Safety AEs of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  AEs will be graded according to the NCI-CTCAE v.5.
Safety Hb of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
Safety neutrophils of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
Safety platelets of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
Safety BT of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
Safety ALT/AST of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
Safety ALK of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
Safety creatinine of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  Parameters Labs will be graded according to the NCI-CTCAE v.5.
QT Assessment | During Day of Cycle 1 (each cycle lasts 21 days)
  The direct relationship between PM534 plasma concentration C and the change from baseline in QT corrected according to Fridericia's formula (ΔQTcF) will be assessed using linear mixed effects (LME) models.
Pharmacokinetics Cmax of PM534 | Cycle 1 from all patients, and also in Cycle 2 from treated patients once the MTD has been determined(each cycle is 21 days).
  Maximum Plasma Concentration (Cmax). Pharmacokinetic analyses will be evaluated in plasma and urine by standard noncompartmental analysis. Compartmental modeling may be performed if appropriate.
Pharmacokinetics AUC of PM534 | Cycle 1 from all patients, and also in Cycle 2 from treated patients once the MTD has been determined(each cycle is 21 days).
  Area Under The Concentration-time Curve (AUC). Pharmacokinetic analyses will be evaluated in plasma and urine by standard noncompartmental analysis. Compartmental modeling may be performed if appropriate.
Pharmacogenomics Plasma AUC(0-t) of PM534 | Cycle 1 from all patients, and also in Cycle 2 from patients treated once the MTD has been determined) (each cycle is 21 days)
  To analyze the expression levels of Plasma AUC(0-t) of response and/or resistance to treatment with PM534
Pharmacogenomics Plasma Cmax of PM534 | Cycle 1 from all patients, and also in Cycle 2 from patients treated once the MTD has been determined) (each cycle is 21 days)
  To analyze the expression levels of Plasma Cmax of response and/or resistance to treatment with PM534
Pharmacogenomics Plasma half life of PM534 | Cycle 1 from all patients, and also in Cycle 2 from patients treated once the MTD has been determined) (each cycle is 21 days)
  To analyze the expression levels of Plasma half life of response and/or resistance to treatment with PM534
Pharmacogenomics Total body plasma clearance of PM534 | Cycle 1 from all patients, and also in Cycle 2 from patients treated once the MTD has been determined) (each cycle is 21 days)
  To analyze the expression levels of Total body plasma clearance of response and/or resistance to treatment with PM534
Pharmacogenomics Volume of distribution of PM534 | Cycle 1 from all patients, and also in Cycle 2 from patients treated once the MTD has been determined) (each cycle is 21 days)
  To analyze the expression levels of Volume of distribution of response and/or resistance to treatment with PM534
Pharmacogenomics Percentage of dose recovered in urine of PM534 | Cycle 1 from all patients, and also in Cycle 2 from patients treated once the MTD has been determined) (each cycle is 21 days)
  To analyze the expression levels of Percentage of dose recovered in urine of response and/or resistance to treatment with PM534
Efficacy of PM534 | From the date of first infusion of PM534 to the date of study termination, up to 46 months
  To analyze the response rates will be determined in patients with measurable or evaluable disease specific tumor types, time-to-event parameter will also be analyzed ORR.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - HM Nou Delfos, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid